CLINICAL TRIAL: NCT06997198
Title: Identification, Assessment, and Treatment of Tardive Dyskinesia With Deutetrabenazine in Adults With Intellectual/Developmental Disabilities and Co-occurring Psychiatric and/or Behavioral Disorders
Brief Title: Deutetrabenazine Treatment for Tardive Dyskinesia in Intellectual/Developmental Disabilities
Acronym: TD-AIDD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, Stephen Ruedrich, Physician, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20250619
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Tardive Dyskinesia; Intellectual Disability; Developmental Disabilities
Keywords: movement disorders; antipsychotic medication adverse effects; Abnormal Involuntary Movement Scale; quality of life; adaptive behavior; caregiver burden; deutetrabenazine; selective vesicular monoamine transporter 2 inhibitor; VMAT2 inhibitor
MeSH Terms: conditions — Tardive Dyskinesia; Intellectual Disability; Developmental Disabilities; Movement Disorders; Caregiver Burden | interventions — deutetrabenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Deutetrabenazine (Experimental): This an open-label study in which all participants will have their Deutetrabenazine dose titrated from 12 mg to 24 mg per day, which will remain the Deutetrabenazine dose through end of study, unless interrupted by adverse events. Participants taking Deutetrabenazine who are concurrently taking strong CYP2D6 inhibitors (paroxetine, fluoxetine, bupropion, duloxetine) will continue their Deutetrabenazine dose at 24 mg per day through end of study.
  Interventions: Drug: Deutetrabenazine Oral Capsule

INTERVENTIONS:
Drug: Deutetrabenazine Oral Capsule — Open-label twenty-four-week treatment with Deutetrabenazine oral tablets (up to 24 mg/day) to test the safety and effectiveness of this medication in ameliorating the signs of tardive dyskinesia in persons with intellectual disability.
  Other Names: Austedo

SUMMARY:
The primary goal of this study is to investigate the efficacy of deutetrabenazine treatment of TD in this previously untreated patient population. Compare movement disorder deutetrabenazine treatment response in persons with IDD to response seen in patients without IDD treated with deutetrabenazine in other treatment settings (per literature review). Compare global deutetrabenazine treatment response with validated instruments.

In addition, we plan to:

* Assess the safety of deutetrabenazine in the treatment of TD in persons with IDD.
* Assess change in Activities of Daily Living (ADLs) in persons with IDD and TD treated with deutetrabenazine, utilizing a validated ADL instrument.
* Assess change in Quality of Life (QOL) in persons with IDD and TD treated with deutetrabenazine, utilizing a validated QOL instrument.
* Assess caregiver burden with a validated caregiver burden instrument.

In this study, 25 participants with IDD and TD will undergo Deutetrabenazine treatment for 24 weeks. The participants will be seen for a total of 5 visits: at baseline, and at follow up visits at 3 weeks, 6 weeks, 12 weeks, and 24 weeks.

This study does not include a comparison group. Therefore, researchers will compare the response of the study participants to deutetrabenazine treatment with those from a previous reported work that resulted in the FDA approval of this medication. This will be an open-label, Phase 4 study.

DETAILED DESCRIPTION:
Tardive dyskinesia (TD) is recognized as a common and often debilitating movement disorder, associated with treatment of a variety of illnesses with dopamine receptor-blocking medications (also commonly known as antipsychotic medications. In addition to the distressing and disfiguring movements of TD, there is now also evidence of reduced quality of life in patients with TD compared to peers with similar psychiatric disorders without TD.

When originally described, TD had been thought to be primarily associated with use of First-Generation Antipsychotics (FGA's, also known as typical antipsychotics), but there are now good studies to suggest that TD is also frequently a result of exposure to Second Generation Antipsychotics (SGA's) as well. Deutetrabenazine, a selective vesicular monoamine transporter 2 inhibitor, is now available to treat the symptoms of TD, with a favorable efficacy and safety profile. This medication offers a treatment option for patients - as well as their caregivers and families - affected by TD.

Individuals with intellectual and developmental disabilities (IDD) commonly suffer from co-occurring psychiatric and/or behavioral disorders (informally known as a "dual diagnosis"). Such individuals are commonly prescribed antipsychotic medications to treat these co-occurring disorders. Several authors have noted that antipsychotic medications have frequently been over-prescribed for individuals with IDD, often in the absence of an identified psychotic illness. Some studies have shown that up to 20-30% of adults with IDD are prescribed antipsychotic medications across a variety of residential settings.

Surrounding this frequent use of antipsychotic medications in persons with IDD, it is now well-established that persons and that having intellectual disability is a recognized risk factor for developing TD when treated with antipsychotic medications. Finally, recent research has confirmed the long-suspected belief that persons with IDD are MORE susceptible to movement disorder side effects when treated with antipsychotic medications when compared to persons without IDD.

Based on their increased exposure to antipsychotics, and increased susceptibility to movement disorders including TD, it would seem that persons with IDD who have TD are a group who could benefit most from treatment with an agent which can address this movement disorder.

Before TD can be treated, it must be clinically identified and formally diagnosed. Once diagnosed, patients and families must be educated on the availability of treatment options, outcomes when no treatment is undertaken, and the potential benefits (and risks) of treatment itself.

Movement disorders such as TD have been diagnosed on the basis of clinical examination, often using formal assessment tools to identify and quantify the movement abnormalities seen. One such instrument is the Abnormal Involuntary Movement Scale (AIMS). The AIMS has been used for many years as the gold standard for this purpose. In addition, there have been recent attempts to quantify the amount of improvement (change in movement intensity, and reduction in AIMS scores) that are considered clinically significant in rating improvement. Additionally, a number of authors have noted the difficulty in using the AIMS in persons with IDD who cannot cooperate fully in the examination process. For this reason, some have suggested using videotaped AIMS exams as a methodology for more accurately quantifying change. Videotaping of exams pre- and post-treatment for blind rating of improvement has been a methodology utilized in a number of recent TD studies.

There is recent initial research attempting to identify and/or quantify the consequence of TD on activities of daily living (ADLs) and quality of life (QOL) of affected individuals; as well as the caregiver burden that may accompany TD for family and non-family caregivers of affected individuals. The Impact-TD scale was developed by TD clinician experts through a modified Delphi process, and produces subscale scores across four domains (social, psychological/psychiatric, physical, vocational/educational/recreational), resulting in a global Impact-TD score. The Impact-TD can utilize input from patients, families, caregivers and clinicians in arriving at subscale and global scores. The Tardive Dyskinesia Impact Scale (TDIS) evolved from a previous scale (the Tardive Dyskinesia Rating Scale) using input from patients and caregivers. The TDIS is an eleven-item questionnaire using a five-point Likert scale to produce a total scale score ranging from 0-44, with higher scores reflecting greater impact of TD on daily functioning. In a small sample of patients with TD, the TDIS appeared valid and reliable. Interestingly, in this sample, TDIS scores did not appear to correlate with AIMS score, indicating that the two scales seemed to capture different aspects of TD severity and consequence.

To date, neither the Impact-TD nor the TDIS have included subjects with IDD and TD. The subjects included in TD studies to date (both the treatment studies of the two VMAT2 inhibitors currently available, and the subsequent studies of the Impact-TD and TDIS) have had diagnoses of schizophrenia, schizoaffective disorder, and mood disorders. Although persons with IDD can and do suffer from these co-occurring psychiatric disorders, this group of individuals have mostly been excluded from TD studies.

The Waisman Activities of Daily Living Scale (W-ADL) is a 17 item instrument rated on a 3-point scale, which has been used in both snapshot and longitudinal studies, and has been shown to have construct validity and few floor or ceiling effects, as well as reliability over time. The World Health Organization Quality of Life Disability Scale (WHO-QOL-D) caregiver form has been used to measure QOL in adults with various disabilities, including intellectual disability. The Zarit Caregiver Burden Scale has been utilized to measure/monitor caregiver burden in individuals with dementia over time. Accordingly, these instruments will be administered pre-and-post treatment of a cohort of adults with ID and TD, in order to determine whether successful treatment of TD will mitigate ADLs and QOL in affected individuals, and caregiver burden in their family and non-family caregivers.

The primary end point of this clinical study is to measure the efficacy of deutetrabenazine in improving TD and reducing AIMS total score. Secondary objectives are to determine whether deutetrabenazine treatment will produce significant improvement in activities of daily living, quality of life; and reduce caregiver burden, in persons with IDD and TD.

ELIGIBILITY:
Participant Inclusion Criteria:

* Diagnosis of IDD (IQ < 70; social/adaptive dysfunction, onset < age 22) as per DSM-5
* Clinical diagnosis of Tardive Dyskinesia (TD) per DSM-5 for at least 3 months before study inclusion (presence of movement disorder for at least 3 months, in absence of previous formal diagnosis of TD).
* Eligible to receive deutetrabenazine, according to current product labeling Stable doses of all psychotropic medications for minimum of three months before study inclusion
* Willing to remain on stable doses of all psychotropics for 24 weeks of study. If female of childbearing age, practicing acceptable form of birth control throughout study duration.
* Subject able to comply with scheduled visits and assessments
* Consent of subject, or legally authorized representative to study protocol.

Caregiver Inclusion Criteria:

* Able to understand and answer questionnaires
* Able to comply with scheduled visits
* Ability to be primary Caregiver for 24 weeks of study

Participant Exclusion Criteria:

* Previous treatment with a VMAT2 inhibitor (tetrabenazine, valbenazine, or deutetrabenazine).
* Treatment with any investigational drug in the 30 days prior to study entry.
* Currently taking a strong CYP2D6 inhibitor such as fluoxetine, paroxetine, quinidine, bupropion. Current treatment with strong anticholinergic agents, monoamine oxidase inhibitors, metoclopramide, dopamine agonists, L-DOPA, or stimulants within past 30 days, or botulinum toxin within the past 3 months.
* Any unstable medical condition in the 60 days prior to study entry.
* Pregnant or breast-feeding
* Current or recent hepatic impairment
* History of neuroleptic malignant syndrome
* History of long QTc on electrocardiogram, bundle branch block (BBB), atrioventricular block, serious cardiac arrhythmia, or heart failure.

QTc on EKG > 450 msec (Fredericia formula) on EKG within 3 months prior to study entry.

* History of substance abuse or dependence in the 3 months prior to study entry.
* Significant risk of suicide or dangerous aggression to others at time of or 3 months prior to study entry.
* Inability to take study medications

Caregiver Exclusion Criteria:

* Unable to complete questionnaires
* Unable to comply with scheduled visits
* Will not be a primary Caregiver for the 24 weeks of the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in AIMS total scores of items 1-7 | Baseline and 24 weeks from start of treatment
  The Abnormal Involuntary Movement Scale (AIMS) has been used for many years as the gold standard for this purpose and the amount of improvement (change in movement intensity, and reduction in AIMS scores) have been assessed clinical significance in rating improvement. A number of authors have noted the difficulty in using the AIMS in persons with IDD who cannot cooperate fully in the examination process. For this reason, some have suggested using videotaped AIMS exams as a methodology for more accurately quantifying change. Videotaping of exams pre- and post-treatment for blind rating of improvement has been a methodology utilized in a number of recent studies of valbenazine. The minimum value of the AIMS total score of items 1-7 is 0 and the maximum value is 49. Higher total AIMS scores mean worse outcomes.

SECONDARY OUTCOMES:
CGI-C | Baseline and 24 weeks from start of treatment
  Clinical Global Impression of Change (CGI-C), as the names indicates, denotes the clinician's impression of change between baseline and after the treatment in which -3 will be marked worsening, -2 moderate worsening, -1 mild worsening, 0 no change, +1 will be marked for mild improvement, +2 moderate improvement, and +3 marked improvement.
CaGI-C | Baseline and 24 weeks from start of treatment
  Caregiver Global Impression of Change (CaGI-C). This is similar to the CGI-C, except that this is the impression of the participant's caregiver, -3 will be marked worsening, -2 moderate worsening, -1 mild worsening, 0 no change, +1 will be marked for mild improvement, +2 moderate improvement, and +3 marked improvement.
Change in ABC-I score | Baseline and 24 weeks from start of treatment
  The Aberrant Behavioral Checklist, Irritability Subscale (ABC-I) is commonly used in clinical trials. It consists of 15 items, which are scored on a 4-point Likert scale of severity, ranging from "not at all a problem" to "the problem is severe in degree."
Change in W-ADL score | Baseline and 24 weeks from start of treatment
  The Waisman Activities of Daily Living (W-ADL) Scale for adolescents and adults with developmental disabilities, is a validated scale that consists of 17 items in the final version of the W-ADL pertain to the current or expected performance of the target individual at the time when the survey was given. The target adult's performance of each activity is rated on a 3-point scale (0 = "does not do at all", 1 = "does with help", 2 = "independent"), and item scores are summed to produce an overall score. Therefore, this means that the scores can range from a minimum of 0 to a maximum value of 51. Higher total W-ADL scores mean better outcomes.
Change in Zarit Burden Interview (short version) score | Baseline and 24 weeks from start of treatment
  The short version of the Zarit Burden Interview is suitable across diagnostic groups of cognitively impaired older adults, and can be used in cross-sectional, longitudinal, and intervention studies. It consists of 12 items, which are answered by a caregiver and measures the change over time, resulting from the progression of (or therapeutic effect of an intervention on) the care recipient's condition. Each item is scored on a 5-point Likert scale, with higher scores indicating greater burden, i.e., worse outcome.
Change in WHOQOL-DIS score | Baseline and 24 weeks from start of treatment
  The World Health Organization Quality of Life Scale- For Persons with Disability (WHOQOL-DIS) is a proxy-reported instrument designed for individuals with either IDD or physical disabilities. It can be used in cross-sectional, longitudinal, and intervention studies. Seventeen items are clustered in four domains: staff quality (4 items), accessibility of care (4 items), meeting needs (5 items), and information (5 items). QOCS for individuals with IDD is scored on a 3-point Likert scales (range 1-3). Total QOCS score are obtained simply by summing the raw individual item scores and converting the sum into score in a 0-100 scale, with higher scores indicating greater quality.
Change in Impact-TD score | Baseline and 24 weeks from start of treatment
  The Impact-TD considers information derived from the participants, caregivers, and clinicians to estimate the level of impact associated with movements due to tardive dyskinesia (TD). For multiple inferences within a domain, the domain score should reflect the highest degree of impact on functioning. Although impact in each domain should be considered, the highest impact in any domain should be considered the single global score. Impact-TD considers the degree of interference, distress, and/or frequency for each of 4 domains (Social, Psychological/ Psychiatric, Physical and Vocational/ Educational/ Recreational). Impact scores in each domain range from 0 to 3, where 0 = no impact, 1 = mild impact (impact is present, but minimal), 2 = moderate impact (exceeds minimal impact, but is not severe), and 3 = severe impact (significant and detrimental impact). Higher scores indicate greater impact, i.e., worse outcome.

OTHER OUTCOMES:
Change Simpson-Angus Scale for EPS | Baseline and 24 weeks from start of treatment
  The Simpson-Angus Scale is a tool used to assess the severity of extrapyramidal symptoms (EPS), which are side effects of antipsychotic medications. The scale consists of ten items that assess five domains: gait, arm dropping, shoulder shaking, elbow rigidity, and wrist rigidity or fixation of position. Each item is rated on a 5-point scale of severity (0 = normal; 4 = most severe; NR = not rated). The total score ranges from 0 to 40, with higher scores indicating more severe EPS outcome.
Change in Barnes Akathisia Scale | Baseline and 24 weeks from start of treatment
  The Barnes Akathisia Scale is a rating scale used to assess the severity of drug-induced akathisia (a syndrome of motor restlessness). It is the most widely used rating scale for akathisia. The scale consists of four items that rate the observable, restless movements that characterize the condition, the subjective awareness of restlessness, and any distress associated with the akathisia. The scale is scored on a 4-point scale from 0-3 and is summed yielding a total score ranging from 0 to 9. The higher the score, the more severe the akathisia, i.e., the worse the outcome.
Assessment of electrocardiogram (EKG)-derived QT/QTc intervals | Baseline and 24 weeks from start of treatment
  QTc intervals have clinical importance as a biomarker of potential drug toxicity. QTc intervals ≥ 450 ms are generally considered long, and drug-induced QTc interval prolongations ≥ 60 ms are generally considered clinically relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ruedrich, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Trial data can be made available on reasonable request to the principal investigator and must be accompanied by detailed study proposals, a description of study objectives, and a statistical analysis plan. Access to available deidentified participant data and the trial protocol may be granted 12 months after publication.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: From 12 months after publication until three years afterwards.
Access Criteria: Any request must be approved by the corresponding author and the principal investigator. Each request will be checked for compatibility with regulatory (institutional review board) requirements as well as compatibility with participant informed consent.

REFERENCES:
- [Background] Townsend-White C, Pham AN, Vassos MV. Review: a systematic review of quality of life measures for people with intellectual disabilities and challenging behaviours. J Intellect Disabil Res. 2012 Mar;56(3):270-84. doi: 10.1111/j.1365-2788.2011.01427.x. Epub 2011 Jun 17. PMID 21679329
- [Background] Tsiouris JA. Pharmacotherapy for aggressive behaviours in persons with intellectual disabilities: treatment or mistreatment? J Intellect Disabil Res. 2010 Jan 1;54(1):1-16. doi: 10.1111/j.1365-2788.2009.01232.x. Epub 2009 Dec 8. PMID 20122096
- [Background] Jain R, Ayyagari R, Goldschmidt D, Zhou M, Finkbeiner S, Leo S. Impact of tardive dyskinesia on patients and caregivers: a survey of caregivers in the United States. J Patient Rep Outcomes. 2023 Nov 28;7(1):122. doi: 10.1186/s41687-023-00658-9. PMID 38015301
- [Background] Jackson R, Brams MN, Carlozzi NE, Citrome L, Fritz NE, Hoberg AR, Isaacson SH, Kane JM, Kumar R. Impact-Tardive Dyskinesia (Impact-TD) Scale: A Clinical Tool to Assess the Impact of Tardive Dyskinesia. J Clin Psychiatry. 2022 Nov 28;84(1):22cs14563. doi: 10.4088/JCP.22cs14563. PMID 36449471
- [Background] Feve A, Angelard B, Lacau St Guily J. Laryngeal tardive dyskinesia. J Neurol. 1995 Jul;242(7):455-9. doi: 10.1007/BF00873549. PMID 7595677
- [Background] Fernandez HH, Factor SA, Hauser RA, Jimenez-Shahed J, Ondo WG, Jarskog LF, Meltzer HY, Woods SW, Bega D, LeDoux MS, Shprecher DR, Davis C, Davis MD, Stamler D, Anderson KE. Randomized controlled trial of deutetrabenazine for tardive dyskinesia: The ARM-TD study. Neurology. 2017 May 23;88(21):2003-2010. doi: 10.1212/WNL.0000000000003960. Epub 2017 Apr 26. PMID 28446646
- [Background] Thurman AJ, Swinehart SS, Klusek J, Roberts JE, Bullard L, Marzan JCB, Brown WT, Abbeduto L. Daily Living Skills in Adolescent and Young Adult Males With Fragile X Syndrome. Am J Intellect Dev Disabil. 2022 Jan 1;127(1):64-83. doi: 10.1352/1944-7558-127.1.64. PMID 34979036
- [Background] Farber RH, Stull DE, Witherspoon B, Evans CJ, Yonan C, Bron M, Dhanda R, Jen E, Brien CO'. The Tardive Dyskinesia Impact Scale (TDIS), a novel patient-reported outcome measure in tardive dyskinesia: development and psychometric validation. J Patient Rep Outcomes. 2024 Jan 4;8(1):2. doi: 10.1186/s41687-023-00679-4. PMID 38175450
- [Background] Anderson KE, Stamler D, Davis MD, Factor SA, Hauser RA, Isojarvi J, Jarskog LF, Jimenez-Shahed J, Kumar R, McEvoy JP, Ochudlo S, Ondo WG, Fernandez HH. Deutetrabenazine for treatment of involuntary movements in patients with tardive dyskinesia (AIM-TD): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Psychiatry. 2017 Aug;4(8):595-604. doi: 10.1016/S2215-0366(17)30236-5. Epub 2017 Jun 28. PMID 28668671
- [Background] Aman MG (2012) Aberrant Behavior Checklist: Current Identity and Future Developments. Clin Exp Pharmacol 2:e114. doi:10.4172/2161- 1459.1000e114
- [Background] Barnes TR. The Barnes Akathisia Rating Scale--revisited. J Psychopharmacol. 2003 Dec;17(4):365-70. doi: 10.1177/0269881103174013. PMID 14870947
- [Background] Bowring DL, Totsika V, Hastings RP, Toogood S, McMahon M. Prevalence of psychotropic medication use and association with challenging behaviour in adults with an intellectual disability. A total population study. J Intellect Disabil Res. 2017 Jun;61(6):604-617. doi: 10.1111/jir.12359. Epub 2017 Jan 16. PMID 28090687
- [Background] Correll CU, Kane JM, Citrome LL. Epidemiology, Prevention, and Assessment of Tardive Dyskinesia and Advances in Treatment. J Clin Psychiatry. 2017 Sep/Oct;78(8):1136-1147. doi: 10.4088/JCP.tv17016ah4c. PMID 29022654
- [Background] de Kuijper GM, Hoekstra PJ. Physicians' reasons not to discontinue long-term used off-label antipsychotic drugs in people with intellectual disability. J Intellect Disabil Res. 2017 Oct;61(10):899-908. doi: 10.1111/jir.12385. Epub 2017 May 30. PMID 28560761
- [Background] de Kuijper GM, Hoekstra PJ. Assessment of Drug-Associated Extrapyramidal Symptoms in People With Intellectual Disability: A Comparison of an Informant-Based Scale With Clinical Rating Scales. J Clin Psychopharmacol. 2016 Oct;36(5):508-12. doi: 10.1097/JCP.0000000000000558. PMID 27529770
- [Background] Fodstad JC, Bamburg JW, Matson JL, Mahan S, Hess JA, Neal D, Holloway J. Tardive dyskinesia and intellectual disability: an examination of demographics and topography in adults with dual diagnosis and atypical antipsychotic use. Res Dev Disabil. 2010 May-Jun;31(3):750-9. doi: 10.1016/j.ridd.2010.01.017. Epub 2010 Mar 5. PMID 20207106
- [Background] Guy W (1976). ECDEU Assessment Manual for Psychopharmacology: Revised (DHEW publication number ADM 76-338). Rockville, MD, Us Department of Health, Education and Welfare, PHS, ADAMHA, NIMH Psychopharmacology Research Branch, Division of Extramural Research Programs, 1976:534-537.
- [Background] Hérbert, R., Bravo, G., & Préville, M. (2000). Reliability, validity, and reference values of the Zarit Burden Interview for assessing informal caregivers of community-dwelling older persons with dementia. Canadian Journal on Aging, 19, 494-507.
- [Background] Kane JM, Correll CU, Nierenberg AA, Caroff SN, Sajatovic M; Tardive Dyskinesia Assessment Working Group. Revisiting the Abnormal Involuntary Movement Scale: Proceedings From the Tardive Dyskinesia Assessment Workshop. J Clin Psychiatry. 2018 May/Jun;79(3):17cs11959. doi: 10.4088/JCP.17cs11959. PMID 29742330
- [Background] Matson JL, Fodstad JC, Neal D, Dempsey T, Rivet TT. Risk factors for tardive dyskinesia in adults with intellectual disability, comorbid psychopathology, and long-term psychotropic use. Res Dev Disabil. 2010 Jan-Feb;31(1):108-16. doi: 10.1016/j.ridd.2009.08.002. Epub 2009 Aug 31. PMID 19720497
- [Background] McEvoy J, Gandhi SK, Rizio AA, Maher S, Kosinski M, Bjorner JB, Carroll B. Effect of tardive dyskinesia on quality of life in patients with bipolar disorder, major depressive disorder, and schizophrenia. Qual Life Res. 2019 Dec;28(12):3303-3312. doi: 10.1007/s11136-019-02269-8. Epub 2019 Aug 21. PMID 31435866
- [Background] Morton RO, Morton LC, Fedora R. Recognition and Treatment of Tardive Dyskinesia in Individuals with Intellectual Disability. Case Rep Psychiatry. 2020 Dec 11;2020:8886980. doi: 10.1155/2020/8886980. eCollection 2020. PMID 33414976
- [Background] Ruedrich SL. (2016). Psychopharmacology. In Hemmings C & Bouras N (eds.) Psychiatric and Behavioural Disorders in Intellectual and Developmental Disabilities, Third Edition, Cambridge University Press, Cambridge, UK, 139-150.
- [Background] Ruedrich SL (2010). Mental Illness in O'Hara J, McCarthy J, and Bouras N. (eds.) Intellectual Disability and Ill Health: A Review of the Evidence, Cambridge University Press, Cambridge UK, 165-177.
- [Background] Ruedrich SL, Diana L, Rossvanes CF, Toliver J. (2005). The abnormal involuntary movement scale (AIMS) and tardive dyskinesia in persons with developmental disability: the benefit of videotaped exams. Mental Health Aspects of Developmental Disabilities 8(3)94-99.
- [Background] Schmidt S, Power M, Green A, Lucas-Carrasco R, Eser E, Dragomirecka E, Fleck M. Self and proxy rating of quality of life in adults with intellectual disabilities: results from the DISQOL study. Res Dev Disabil. 2010 Sep-Oct;31(5):1015-26. doi: 10.1016/j.ridd.2010.04.013. Epub 2010 May 15. PMID 20478692
- [Background] Schooler NR, Kane JM. Research diagnoses for tardive dyskinesia. Arch Gen Psychiatry. 1982 Apr;39(4):486-7. doi: 10.1001/archpsyc.1982.04290040080014. No abstract available. PMID 6121550
- [Background] Sheehan R, Horsfall L, Strydom A, Osborn D, Walters K, Hassiotis A. Movement side effects of antipsychotic drugs in adults with and without intellectual disability: UK population-based cohort study. BMJ Open. 2017 Aug 3;7(8):e017406. doi: 10.1136/bmjopen-2017-017406. PMID 28775195
- [Background] Simpson GM, Angus JW. A rating scale for extrapyramidal side effects. Acta Psychiatr Scand Suppl. 1970;212:11-9. doi: 10.1111/j.1600-0447.1970.tb02066.x. No abstract available. PMID 4917967
- [Background] Solmi M, Pigato G, Kane JM, Correll CU. Clinical risk factors for the development of tardive dyskinesia. J Neurol Sci. 2018 Jun 15;389:21-27. doi: 10.1016/j.jns.2018.02.012. Epub 2018 Feb 5. PMID 29439776
- [Background] Stacy M, Sajatovic M, Kane JM, Cutler AJ, Liang GS, O'Brien CF, Correll CU. Abnormal involuntary movement scale in tardive dyskinesia: Minimal clinically important difference. Mov Disord. 2019 Aug;34(8):1203-1209. doi: 10.1002/mds.27769. Epub 2019 Jun 24. PMID 31234240
- [Background] Whiteney C and Evered JA (2022). The Qualitative Research Distress Protocol: A Participant-Centered Tool for Navigating Distress During Data Collection. International Journal of Qualitative Methods Volume 21:1-9.
- [Background] Woods SW, Morgenstern H, Saksa JR, Walsh BC, Sullivan MC, Money R, Hawkins KA, Gueorguieva RV, Glazer WM. Incidence of tardive dyskinesia with atypical versus conventional antipsychotic medications: a prospective cohort study. J Clin Psychiatry. 2010 Apr;71(4):463-74. doi: 10.4088/JCP.07m03890yel. Epub 2010 Feb 9. PMID 20156410
- [Background] Yu J, Yap P, Liew TM. The optimal short version of the Zarit Burden Interview for dementia caregivers: diagnostic utility and externally validated cutoffs. Aging Ment Health. 2019 Jun;23(6):706-710. doi: 10.1080/13607863.2018.1450841. Epub 2018 Mar 19. PMID 29553806